CLINICAL TRIAL: NCT02917733
Title: Disposition of [¹⁴C₂]-Labeled LY3039478 Following Oral Administration in Healthy Subjects
Brief Title: A Study of the Absorption, Distribution, Metabolism and Excretion of LY3039478 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 16343; I6F-MC-JJCF (Other: Eli Lilly and Company)
Record Dates: First submitted 2016-09-15; First posted 2016-09-28 (Estimated); Results first posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Healthy
MeSH Terms: interventions — crenigacestat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Radiolabelled LY3039478 (Experimental): Single dose of radiolabelled LY3039478 administered orally.
  Interventions: Drug: LY3039478

INTERVENTIONS:
Drug: LY3039478 — Administered orally

SUMMARY:
This type of study is called a radiolabeled study. For this study, LY3039478 (study drug) has been specially prepared to contain radiolabeled carbon [¹⁴C]. [¹⁴C] is a naturally occurring radioactive form of the element carbon. This study will help determine how the drug appears in the blood, urine, and stool after it is administered by mouth to healthy people. Information about any side effects that may occur will also be collected. This study will last about 10 weeks for each participant.

ELIGIBILITY:
Inclusion Criteria:

- Have a body mass index (BMI) of 18 to 32 kilogram per meter square (kg/m²), inclusive

Exclusion Criteria:

* Have previously completed or withdrawn from this study or any other study investigating LY3039478, and have previously received the investigational product
* Have known allergies to LY3039478, related compounds or any components of the formulation, or history of significant atopy
* Have had exposure to significant diagnostic, therapeutic, or employment-related radiation within 12 months prior to dosing (eg, serial x-ray or computed tomography scans, barium meal, current employment in a job requiring radiation exposure monitoring)
* Have participated in a [¹⁴C] study within the last 6 months prior to admission for this study. The total 12-month exposure from this study and a maximum of one other previous [¹⁴C]-study within 6 to 12 months of this study must be within the Code of Federal Regulations (CFR) recommended levels considered safe: less than 5000 millirem (mrem)/year whole body annual exposure

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-09; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Covance Clinical Research Inc, Madison, Wisconsin, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- 75 mg [14C2] LY3039478: Participants received approximately 75 mg [14C2] LY3039478 containing approximately 100 μCi [14C2] LY3039478.
Period: Overall Study
Arm/Group | 75 mg [14C2] LY3039478
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All participants who received the [14C2]-LY3039478 dose.
Arm/Group | 75 mg [14C2] LY3039478
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.0 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Urinary and Fecal Excretion of Radioactivity Over Time Expressed as a Percentage of the Total Radioactive Dose Administered
Description: To determine the disposition of radioactivity and LY3039478 in healthy participants following oral administration of a single dose 14C-labeled LY3039478.
Time Frame: Predose, and at 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48, 72, 96, 120, 144, 168, 192, 216, 240, 264, 288, and 312 hours postdose
Population: All participants who received the [14C2]-LY3039478 dose.
Measure: Mean (Standard Deviation); unit: percentage of administered radioactivity
Arm/Group | 75 mg [14C2] LY3039478
Number analyzed (Participants) | 6
percentage of administered radioactivity | 90.2 (2.32)

2. Secondary Outcome: Pharmacokinetics: Area Under the Concentration Versus Time Curve From Time Zero to Infinity (AUC[0-inf]) of LY3039478
Description: The AUC[0-inf]) for plasma LY3039478 was evaluated by using a combination of the linear and logarithmic trapezoidal methods (linear-log trapezoidal rule).
Time Frame: Predose, and at 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48, 72, 96, 120, 144, and 168 hours postdose
Population: All the participants who received [14C2]-LY3039478 dose and had evaluable data for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hour/milliliter (ng*h/mL)
Arm/Group | 75 mg [14C2] LY3039478
Number analyzed (Participants) | 5
nanograms*hour/milliliter (ng*h/mL) | 2570 (11)

3. Secondary Outcome: Pharmacokinetics: Area Under the Concentration Versus Time Curve From Time Zero to Infinity (AUC[0-inf]) of Total Plasma Radioactivity
Description: The AUC[0-inf]) for total plasma radioactivity was evaluated by using a combination of the linear and logarithmic trapezoidal methods (linear-log trapezoidal rule).
Time Frame: Predose, and at 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48, 72, 96, 120, 144, and 168 hours postdose
Population: All the participants who received [14C2]-LY3039478 dose and had evaluable data for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng quivalents*hour/gram (ng equiv.h/g)
Arm/Group | 75 mg [14C2] LY3039478
Number analyzed (Participants) | 4
ng quivalents*hour/gram (ng equiv.h/g) | 26100 (21)

4. Secondary Outcome: Pharmacokinetics: Maximum Observed Concentration (Cmax) of LY3039478
Description: The Cmax of LY3039478 was evaluated.
Time Frame: Predose, and at 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48, 72, 96, 120, 144, and 168 hours postdose
Population: All the participants who received [14C2]-LY3039478 dose and had evaluable data for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms/milliliter (ng/ml)
Arm/Group | 75 mg [14C2] LY3039478
Number analyzed (Participants) | 5
Nanograms/milliliter (ng/ml) | 517 (15)

5. Secondary Outcome: Pharmacokinetics: Maximum Observed Concentration (Cmax) of Total Plasma Radioactivity
Description: Cmax of total plasma radioactivity was evaluated.
Time Frame: Predose, and at 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48, 72, 96, 120, 144, and 168 hours postdose
Population: All participants who received [14C2]-LY3039478 dose and had evaluable data for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms equivalents/gram (ng equiv/g)
Arm/Group | 75 mg [14C2] LY3039478
Number analyzed (Participants) | 5
Nanograms equivalents/gram (ng equiv/g) | 1060 (10)

6. Secondary Outcome: Total Number of Metabolites of LY3039478 in Plasma, Urine and Feces
Description: Following oral administration, radio high performance liquid chromatography (HPLC) and liquid chromatography-mass spectrometry (LC-MS) profiles were obtained from analysis of plasma, urine and feces.
Time Frame: Predose, and at 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48, 72, 96, 120, 144, and 168 hours postdose.
Population: All participants who received [14C2]-LY3039478 dose. For the feces profiling, only one participant had quantifiable radioactive dose recovered in feces adequate for metabolite profiling and was therefore eligible for analysis.
Measure: Number; unit: Metabolites
Arm/Group | 75 mg [14C2] LY3039478
Number analyzed (Participants) | 6
Metabolites
  Number of Metabolites of LY3039478 in Plasma | 8
  Number of Metabolites of LY3039478 in Urine | 10
  Number of Metabolites of LY3039478 in Feces: number analyzed (Participants) | 1
  Number of Metabolites of LY3039478 in Feces | 3

ADVERSE EVENTS:
Description: All the participants who received the [14C2]-LY3039478 dose.
Groups:
- 75 mg [14C2] LY3039478: All the participants received approximately 75 mg [14C2] LY3039478 containing approximately 100 μCi [14C2] LY3039478, with the exception of participant 01005 who received a lower than expected dose (84.5249 µCi, rather than the target dose of 100 µCi).
Arm/Group | 75 mg [14C2] LY3039478
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 6/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 75 mg [14C2] LY3039478 (N=6)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2)
Haematochezia (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Fatigue (General disorders) | 2 (2)
Feeling hot (General disorders) | 1 (1)
Scratch (Injury, poisoning and procedural complications) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Presyncope (Nervous system disorders) | 1 (1)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less